CLINICAL TRIAL: NCT05083884
Title: Prospective Survey of Women With Vasomotor Symptoms Associated With Menopause in Nordic Europe, Canada, Brazil and Mexico - WARM Study
Brief Title: A Survey About Hot Flashes in Women Going Through the Menopause
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 2693-MA-3235
Record Dates: First submitted 2021-10-07; First posted 2021-10-19 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Menopause; Vasomotor Symptoms
Keywords: Menopause; Vasomotor Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Peri-menopausal woman: Grouping is based on Peri-menopausal woman
  Interventions: Other: No Intervention
- Group 2: Post- menopausal woman: Grouping is based on Post-menopausal woman
  Interventions: Other: No Intervention
- Group 3: Peri-menopausal woman: moderate-to-severe MR-VMS: Grouping is based on Peri-menopausal woman with moderate-to-severe vasomotor symptoms (MR-VMS)
  Interventions: Other: No Intervention
- Group 4: Post-menopausal woman: moderate-to-severe MR-VMS: Grouping is based on Post-menopausal woman with moderate-to-severe vasomotor symptoms (MR-VMS)
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a cross-sectional non-product related survey including peri- and post-menopausal women with moderate to severe VMS associated with menopause.

SUMMARY:
This study is an online survey of women in and around menopause with moderate to severe hot flashes. Menopause, a normal part of life, is a time after a woman's last period. Hot flashes often occur during menopause. They can disrupt a woman's daily life.

This study is about collecting information only. There will be no treatment in this study.

This study will provide information about how many women have moderate to severe hot flashes in menopause. It will also provide details on women's experiences with hot flashes.

Women from Brazil, Canada, Nordic Europe, and Mexico will take part in this study. The women in this study will already be taking part in consumer panels. Women will be contacted based on their age. They will be asked if they would like to take part in this study.

Firstly, the women will answer questions about whether they are in menopause or are getting close to menopause. They will also be asked how severe their hot flashes are.

From their answers, some women will be asked to complete an online survey. These will be women who are in menopause and have moderate to severe hot flashes. They will provide more details about how hot flashes have impacted their lives. Also, they will answer questions on how hot flashes affect their quality of life. Finally, they will answer questions about their experiences when they visited their doctor about their hot flashes.

ELIGIBILITY:
Inclusion Criteria (primary outcome measure):

- Post-menopausal women

Inclusion Criteria (secondary outcome measure):

* Women currently experiencing, or have experienced in the last month, moderate to severe VMS symptoms (i.e. minimum of 1 moderate to severe hot flushes per day over the last month)
* Peri-menopausal and post-menopausal women

Exclusion Criteria (primary outcome measure):

* Women with current breast cancer treatment
* Women treated with anti-estrogens, aromatase inhibitors or Gonadotropin-releasing hormone (GnRH) agonists/antagonists for cancer or any other medical condition.

Additional exclusion criterion for secondary outcome measures will be:

- Mild VMS symptoms only

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Peri- and post-menopausal women with moderate to severe VMS symptoms
Sampling Method: Non-Probability Sample
Enrollment: 2176 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
Prevalence of moderate to severe vasomotor symptoms (VMS) in post-menopausal women | 1 day (once through survey)
  Prevalence of moderate to severe VMS in post-menopausal women. Post-menopause is defined as at least 12 consecutive months without a period. Moderate VMS associated with menopause symptoms is defined as sensations of heat with sweating but being able to continue activities. Severe VMS associated with menopause is defined as feelings of intense heat with sweating causing cessation of activities. The recall period is 1 month prior to survey.

SECONDARY OUTCOMES:
Health Related Quality of Life (HRQoL) measured by the Menopause Specific QoL Questionnaire (MENQoL) | 1 day (once through survey)
  MENQoL measures the overall score and four domain-specific scores assessing wellbeing (vasomotor; psychosocial; physical; sexual). Scores range from 1 to 8 with a higher score indicating worsening/increasing bothersomeness by the symptom experience. The MENQoL recall period is 7 days prior to survey.
Health Related Quality of Life (HRQoL) measured by Work Productivity and Activity Impairment-VMS (WPAI-VMS) Questionnaire | 1 day (once through survey)
  The WPAI-VMS questionnaire measures four domain specific scores assessing work productivity and activity impairment over the previous week (absenteeism; presenteeism; mean work productivity; activity impairment). Scores range from 0 to 100%. The four scores were expressed as impairment percentages with a higher score indicating less productivity and greater activity impairment. The WPAI recall period is 7 days prior to survey.
Health Related Quality of Life (HRQoL) measured by Patient-Reported Outcomes Measurement Information System - Sleep Disturbance (PROMIS) | 1 day (once through survey)
  The PROMIS Sleep Disturbance instrument assesses self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep. Each item on the measure is rated on a 5-point scale with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance. The PROMIS recall period is 7 days prior to survey.
  (Only implemented in Canada, Brazil and Denmark).
Proportion of Participants with VMS seeking healthcare professionals' (HCP) advice | 1 day (once through survey)
  The type of specialists reported by peri- and post-menopausal women will be assessed.
Proportion of Participants with VMS taking over the counter treatment for moderate to severe VMS symptoms | 1 day (once through survey)
  The types of over the counter treatment taken by peri- and post-menopausal women for MR symptoms will be assessed.
Proportion of Participants incurring average out-of-pocket expenses incurred in treatment of menopause | 1 day (once through survey)
  Average out-of-pocket expenses incurred in the treatment of menopause reported by medications bought will be assessed.
Percentage of peri-and post-menopausal women who seek help from HCPs for their menopause related symptoms (MR-VMS) | 1 day (once through survey)
  Percentage of peri- and post-menopausal women who seek help from Health Care Professionals (HCPs) for their MR-VMS. Help from an HCP can be in the form of advice or receipt of pharmaceutical treatment.
Health Related Quality of Life (HRQoL) measured by participants' attitudes to their VMS | 1 day (once through survey)
  Participants' attitudes towards their VMS will be evaluated using the following: agreement or disagreement to statements on menopause itself, available treatments, and willingness/aversion to hormone replacement therapy (HRT).
Treatment patterns of peri- and post-menopausal women assessed by type of treatment | 1 day (once through survey)
  The number of peri- and post-menopausal women treated with hormonal treatment, non-hormonal treatment, or other approaches will be summarized.
Treatment patterns of peri- and post-menopausal assessed by length of time on hormonal treatment | 1 day (once through survey)
  The length of time on hormonal treatment in peri- and post-menopausal women will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Medical Affairs Europe
Locations (1):
- IQVIA, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Todorova L, Bonassi R, Guerrero Carreno FJ, Hirschberg AL, Yuksel N, Rea C, Scrine L, Kim JS. Prevalence and impact of vasomotor symptoms due to menopause among women in Brazil, Canada, Mexico, and Nordic Europe: a cross-sectional survey. Menopause. 2023 Dec 1;30(12):1179-1189. doi: 10.1097/GME.0000000000002265. Epub 2023 Oct 19. PMID 37847872
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/2693-MA-3235/